CLINICAL TRIAL: NCT03545763
Title: Evaluating Control of Hypertension - Effect of Social Determinants
Acronym: ECHOES
Status: Completed | Type: Observational
Sponsor: Oregon Health and Science University (Other)
Collaborators: OCHIN, Inc. (Other); National Institutes of Health (NIH) (NIH); National Heart, Lung, and Blood Institute (NHLBI) (NIH); Health Choice Network (Other); Fenway Community Health (Other)
Responsible Party: Principal Investigator, Jennifer E DeVoe, MD DPhil, Chair of the Department of Family Medicine, Oregon Health and Science University
Other Study IDs: R01HL136575 (NIH); R01HL136575 (NIH)
Record Dates: First submitted 2018-05-22; First posted 2018-06-04 (Actual); Last update posted 2024-04-18 (Actual); Status verified 2024-04

CONDITIONS: Hypertension
Keywords: Hypertension; Social Determinants of Health; Health Insurance; Medicaid; Affordable Care Act
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Medicaid Expansion States: Patients receiving care in community health centers in states that expanded Medicaid (intervention group)
  Interventions: Other: Medicaid Expansion
- Non Medicaid Expansion States: Patients receiving care in community health centers in states that did not expand Medicaid (control group)
  Interventions: Other: Medicaid Expansion

INTERVENTIONS:
Other: Medicaid Expansion — There will be no direct intervention, but rather an observation of change based on whether a state expanded Medicaid or not

SUMMARY:
This study evaluates the impact of a large-scale, national expansion of Medicaid on hypertension incidence, screening, treatment, and management. Social Determinants of Health will be assessed as moderators, and comparing states that did versus states that did not expand Medicaid will also be evaluated.

DETAILED DESCRIPTION:
The Affordable Care Act (ACA) enacted several provisions intended to improve healthcare for vulnerable populations,including expanding Medicaid eligibility to those earning ≤138% of the federal poverty level (FPL). Since the expansion was not required, as of March 2018, 32 states (and District of Columbia) implemented the expansion and 18 did not. Simulated models predicted the ACA would improve health outcomes and reduce disparities for patients with hypertension, yet actual changes are not yet available. In addition, there is new interest in tracking and utilizing Social Determinants of Health (SDH) in the primary care setting but there is currently little information on how this information will impact Hypertension (HTN) care, especially related to changes to health insurance availability. This study will build on current understanding of how health insurance impacts HTN incidence, screening, treatment, and management by comparing states that did versus did not expand Medicaid as part of the ACA and seeks to understand the influence of SDH on these changes. the investigators will address the following specific aims: Aim 1: Compare HTN incidence, prevalence of undiagnosed HTN, and rates of HTN screening, in Medicaid expansion versus non-expansion states before and after the ACA. Aim 2: Compare HTN treatment (e.g., medication use), and management (e.g., HTN control, systolic and diastolic blood pressure change, risk factors related to HTN control) in Medicaid expansion versus non-expansion states before and after the ACA. Aim 3: Assess the extent to which rates of HTN incidence, screening, and treatment effectiveness among patients who gained insurance versus those continuously insured or uninsured, pre-post ACA, are moderated by individual-level SDH (e.g., race, ethnicity), in expansion states. Aim 4: Explore the interaction between community-level SDH (e.g., neighborhood racial segregation and deprivation) and HTN incidence, screening, treatment, and management among patients who gained insurance relative to those who were continuously insured or uninsured, in expansion states. The findings from this project will be extremely relevant to policy and practice, informing further improvements in the US healthcare system to ensure access to healthcare for vulnerable populations.

ELIGIBILITY:
Inclusion Criteria:

* Patients in intervention and control states aged 19-64

Exclusion Criteria:

* Patients outside of age range 19-64

Ages: 19 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Study eligible patients within electronic health record data from the Accelerating Data Value Across a National Community Health Center Network (ADVANCE) community health information network
Sampling Method: Non-Probability Sample
Enrollment: 1939783 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2023-04-01 (Actual); Study Completion 2023-05-15 (Actual)

PRIMARY OUTCOMES:
Hypertension incidence | 24 months prior to Medicaid expansion vs 24 months post
  Rates of hypertension diagnosis using the following codes in the EHR: ICD-9: 401.00-401.99, 402.00-405.99 or ICD-10: I10-I15.
Undiagnosed hypertension | 24 months prior to Medicaid expansion vs 24 months post
  high blood pressure but no diagnosis or medications can be noted in the EHR diagnostic codes that can be used to document why a diagnosis of hypertension was not made including ICD-10 R03.0 (i.e., white coat syndrome without HTN) and ICD-9 796.2 (i.e., elevated BP without HTN).
Hypertension screening | 24 months prior to Medicaid expansion vs 24 months post
  rate of blood pressure screening marked in EHR
Hypertension treatment | 24 months prior to Medicaid expansion vs 24 months post
  the number of anti-hypertensive medications prescribed in EHR
Hypertension management | 24 months prior to Medicaid expansion vs 24 months post
  blood pressure control: last measure within range of normal for age/risk(s); percent Y/N at last visit, value/date of last measure

SECONDARY OUTCOMES:
Insurance status and rates of coverage | 24 months prior to Medicaid expansion vs 24 months post
  Health insurance status derived from EHR data and is primarily based on information collected at each visit
Service Utilization | 24 months prior to Medicaid expansion vs 24 months post
  Type of internal services utilized including number and ratio of "traditional" face to face visits vs. "nontraditional" encounters and communication via phone, personal health record, and email
Preventive service receipt | 24 months prior to Medicaid expansion vs 24 months post
  number of all billed encounters overall and yearly, as well as number of cancer screening, smoking screening, lipid screening, diabetes screening, obesity screening
Hypertension related complications | 24 months prior to Medicaid expansion vs 24 months post
  incidence of related complications and diseases derived from EHR data

CONTACTS AND LOCATIONS:
Locations (1):
- Oregon Health & Science University, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Huguet N, Larson A, Angier H, Marino M, Green BB, Moreno L, DeVoe JE. Rates of Undiagnosed Hypertension and Diagnosed Hypertension Without Anti-hypertensive Medication Following the Affordable Care Act. Am J Hypertens. 2021 Sep 22;34(9):989-998. doi: 10.1093/ajh/hpab069. PMID 33929496
- [Derived] Angier H, Huguet N, Marino M, Green B, Holderness H, Gold R, Hoopes M, DeVoe J. Observational study protocol for evaluating control of hypertension and the effects of social determinants. BMJ Open. 2019 Mar 15;9(3):e025975. doi: 10.1136/bmjopen-2018-025975. PMID 30878987